CLINICAL TRIAL: NCT03591627
Title: Left Atrial Thrombus on Transesophageal Echocardiography
Acronym: LATTEE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Agnieszka Kaplon-Cieslicka, Agnieszka Kapłoń-Cieślicka, Medical University of Warsaw, Medical University of Warsaw
Other Study IDs: 1st Department of Cardiology
Record Dates: First submitted 2018-07-07; First posted 2018-07-19 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Transesophageal Echocardiography; Ablation; Cardioversion; Thrombus; Embolism
Keywords: Atrial fibrillation; Atrial Flutter; Transesophageal echocardiography; Ablation; Cardioversion; Thrombus; Embolism
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Thromboembolism | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AF or AFl patients: Patients with AF or AFl in whom TEE will be performed (to assess their eligibility for cardioversion or ablation), hospitalized in a participating center during study period.
  Interventions: Diagnostic Test: Transesophageal echocardiography

INTERVENTIONS:
Diagnostic Test: Transesophageal echocardiography — Transesophageal echocardiography will be used to exclude the presence of an LA thrombus before AF/AFI ablation or cardioversion.

SUMMARY:
The aim of the study is to assess the prevalence of left atrial thrombus in patients with atrial fibrillation (AF) or atrial flutter (AFI), in whom transesophageal echocardiography is performed before AF/AFl cardioversion or ablation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) and atrial flutter (AFI) increase the risk of thromboembolic events by promoting clot formation in the left atrium (LA). Transesophageal echocardiography (TEE) is routinely used to exclude the presence of an LA thrombus before AF/AFI ablation or cardioversion. So far, it has not been established what is the optimal combination of noninvasive parameters for thromboembolic risk stratification in this setting. The present study is aimed to compare the prevalence of LA thrombus in patients on different anticoagulant regimens, identify predictors of LA thrombus and validate the newly developed CHA2DS2-VASc-AF-GFR score (and to compare its predictive value in LA thrombus identification with those of the CHA2DS2-VASc and the CHADS2 scores).

The study protocol all patients with AF or AFl in whom TEE will be performed (to assess their eligibility for cardioversion or ablation), hospitalized in a participating center during study period.

ELIGIBILITY:
Inclusion Criteria:

* All patients with AF or AFl in whom TEE will be performed (to assess their eligibility for cardioversion or ablation), hospitalized in a participating center during study period.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with AF or AFl in whom TEE will be performed (to assess their eligibility for cardioversion or ablation), hospitalized in a participating center during study period.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the prevalence of LA thrombus in patients with AF/AFI, in whom TEE is performed before AF/AFl cardioversion or ablation. | One day

SECONDARY OUTCOMES:
Comparison of the prevalence of LA thrombus in patients on different anticoagulant regimens. | Up to 12 months
Identification of the predictors of LA thrombus. | Up to 12 months
Validation of the the newly developed CHA2DS2-VASc-AF-GFR score (and to compare its predictive value in LA thrombus identification with those of the CHA2DS2-VASc and the CHADS2 scores). | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- 1st Department of Cariology of Medcial University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided